CLINICAL TRIAL: NCT01678690
Title: An Open-Label, Exploratory, Limited Dose Escalation Study to Evaluate the Pharmacokinetics, Safety and Tolerability of Gemcitabine Hydrochloride Oral Formulation (D07001-F4) in Subjects With Malignant Tumors
Brief Title: An Exploratory Study of Gemcitabine Hydrochloride Oral Formulation (D07001-F4) in Subjects With Malignant Tumors
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: InnoPharmax Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: HR-11-001
Record Dates: First submitted 2012-08-29; First posted 2012-09-05 (Estimated); Last update posted 2016-09-02 (Estimated); Status verified 2016-08

CONDITIONS: Malignant Tumors
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gemcitabine HCl Oral Formulation (Experimental): Subjects will be treated with Gemcitabine HCl Oral Formulation according to assigned cohort (2 mg or 5 mg or 10 mg) on Day 1 of the 7-day study treatment period
  Interventions: Drug: Gemcitabine HCl Oral Formulation

INTERVENTIONS:
Drug: Gemcitabine HCl Oral Formulation — Gemcitabine HCl Oral Formulation 80 mg/vial Subjects will be treated on Day 1 of the 7-day study treatment period
  Other Names: D07001-F4

SUMMARY:
Open-label, Phase 0, dose-escalation study of 3 successive cohorts (3 subjects per cohort), to determine and characterize the plasma PK of gemcitabine HCl oral formulation (D07001-F4) administered once on Day 1 with 7 Days of study follow-up. In addition, oral tolerability and safety will also be assessed during this 1-week period.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged 18 years and older.
2. Signed and dated informed consent form.
3. Subjects with malignancies with histological or pathologic confirmation and who are clinically stable.
4. History of treatment with at least 1 cytotoxic chemotherapy regimen for the current malignancy.
5. If the subject has received cytotoxic chemotherapy within the past 14 days, the subject is beyond the nadir of white blood cell and platelet counts.
6. At least 28 days have elapsed since the subject's prior radiotherapy or any major surgery (excluding diagnostic biopsy or venous access device placement).
7. World Health Organization (WHO) performance status 0 to 2
8. Subject has an ANC ≥1500 cells/mm³, platelet count ≥ 100,000 cells/mm³, and hemoglobin ≥ 9 g/dL.
9. Subject has adequate liver function demonstrated by transaminases within normal limits (aspartate transaminase and alanine transaminase), total bilirubin ≤ 1.5 mg/dL (unless due to Gilbert's syndrome), albumin ≥ 2.5 g/dL, international normalized ratio [INR] < 1.5).
10. Subject has adequate renal function: serum creatinine ≤ 1.5 x upper limit of normal.
11. Subject has a life expectancy >24 weeks.
12. If a women of child-bearing potential, subject has a negative pregnancy test and is not breast-feeding.
13. If a women of child-bearing potential, subject is using a medically acceptable form of birth control prior to screening and for the duration of their study participation and for 1 month after the end of the study.
14. Subject is willing to comply with protocol-required visit schedule and visit requirements and provide written informed consent.

Exclusion Criteria:

1. Subject has rapidly progressive disease or rapid clinical deterioration as assessed by the Investigator.
2. Subject is receiving full-dose (therapeutic) anticoagulation therapy.
3. Subject is receiving concomitant radiotherapy.
4. Subject is intolerant or allergic or has a known hypersensitivity to gemcitabine.
5. Subject has clinically significant cardiovascular disease (for example: uncontrolled hypertension, unstable angina, congestive heart failure, or New York Heart Association Grade 2 or greater).
6. Subject has uncontrolled serious cardiac arrhythmia.
7. Subject has known active brain metastases, or any leptomeningeal metastases.
8. Subject has a history of drug or alcohol abuse within last year.
9. Subject has documented cerebrovascular disease.
10. Subject has a seizure disorder not controlled on medication.
11. Subject received an investigational agent within 30 days of screening.
12. Subject received systemic treatment for infection within 14 days of screening.
13. Subject has known human immunodeficiency virus infection or viral hepatitis.
14. Subject has any other serious medical condition that, in the investigator's medical opinion, would preclude safe participation in a clinical trial.
15. Subject has gastrointestinal disease or prior gastrointestinal surgery that may interfere with adequate oral therapy absorption.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2012-08; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
gemcitabine (dFdC) and difluorodeoxyuridine (dFdU) plasma concentration and gemcitabine triphosphate (dFdCTP) concentration in PBMC | Day 1-5

SECONDARY OUTCOMES:
the proportion of subjects experiencing adverse events all grades, change from baseline in clinical laboratory test results, vital sign measurements, and physical examination findings | Day 1-8 (+/- 1) days

CONTACTS AND LOCATIONS:
Overall Officials: Nashat Y. Gabrail, MD, Principal Investigator — Gabrail Cancer Center Research; Sharad Ghamande, MD, Principal Investigator — Augusta University; Chia-Chi Lin, MD, Principal Investigator — National Taiwan University Hospital
Locations (4):
- United States (3):
  - Georgia Regents University- Cancer Center, Augusta, Georgia
  - Gabrail Cancer Center Research, Canton, Ohio
  - Gabrail Cancer Center Research, Dover, Ohio
- National Taiwan University Hospital, Taipei, Taiwan, Taiwan